CLINICAL TRIAL: NCT06435130
Title: The Impact of Chokeberry Bioproducts Consumption on Metabolic Parameters and the Antioxidant Potential of Serum
Brief Title: The Impact of Chokeberry Bioproducts on Metabolic Parameters and Antioxidant Potential
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Małgorzata Zujko, Principal Investigator, Medical University of Bialystok
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MUBialystok2
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diet, Healthy; Diabetes Mellitus; Hypertension; Obesity; Hypercholesterolemia
Keywords: chokeberry; juice; fiber; diet; intervention; diabetes; obesity; hypertension; hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Obesity; Hypercholesterolemia | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: 102 people (67 women and 35 men) with metabolic disorders were included in the interventional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention with chokeberry juice and fibre (Experimental): Study participants consumed 100 mL of chokeberry juice daily for 8 weeks. After 8 weeks, participants consumed 100 ml of chokeberry juice and 10 g of chokeberry fiber daily for 4 weeks.
  Interventions: Other: Dietary intervention with chokeberry juices; Other: Dietary intervention with chokeberry juices and fibers

INTERVENTIONS:
Other: Dietary intervention with chokeberry juices — The first stage of the dietary intervention lasted 8 weeks. Study participants consumed 100 ml of chokeberry juice daily. Chokeberry juice came from ecological cultivation (Poland). Participants qualified for the study had specific biochemical parameters tested: fasting glucose and insulin level, lipid profile (triglycerides, total cholesterol, LDL-cholesterol, HDL-cholesterol), glycated hemoglobin, uric acid, C-reactive protein (CRP), creatinine, liver enzymes: alanine transaminase (ALT), aspartate transaminase (AST), gamma-glutamylotranspeptydase (GGTP), homocysteine and antioxidant potential. Blood tests were performed in a certified external laboratory before and after 8 weeks of intervention. In addition, blood pressure and waist circumference were tested.
Other: Dietary intervention with chokeberry juices and fibers — The second stage of the dietary intervention lasted 4 weeks. Study participants consumed 100 ml of chokeberry juice daily and 10 g chokeberry fiber daily (from ecological cultivation, Poland). Blood tests were performed in a certified external laboratory after 4 weeks of intervention. The following blood tests were performed: fasting glucose and insulin level, lipid profile (triglycerides, total cholesterol, LDL-cholesterol, HDL-cholesterol), glycated hemoglobin, uric acid, C-reactive protein (CRP), creatinine, liver enzymes: alanine transaminase (ALT), aspartate transaminase (AST), gamma-glutamylotranspeptydase (GGTP), homocysteine and antioxidant potential. In addition, blood pressure and waist circumference were tested.

SUMMARY:
Chokeberry can be used both in the prevention and treatment of various metabolic disorders due to its high antioxidant properties. The study assessed for the first time the synergistic effect of chokeberry juice and chokeberry fiber on selected metabolic and anthropometric parameters. 102 people (67 women and 35 men) took part in the intervention study. After 8 weeks of intervention with chokeberry juice and another 4 weeks of intervention with chokeberry juice and fiber, a change in waist circumference, blood pressure, glucose, glycated hemoglobin, LDL cholesterol, aspartate transaminase (AST) and the level of antioxidant potential was observed.

ELIGIBILITY:
Inclusion Criteria:

* age 30-65 years,
* low or moderate physical activity.

Exclusion Criteria:

* age <30 and >65 years,
* high physical activity,
* obesity (class II),
* diabetes (all types),
* gastric ulcer,
* acute or chronic gastritis,
* intestinal diseases, including inflammatory bowel diseases and functional intestinal disorders,
* taking hypoglycemic, lipid-lowering, immunosuppressive, anticoagulant and antihypertensive drugs, use of steroid therapy,
* high physical activity,
* pregnancy,
* breastfeeding.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in waist circumference | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in waist circumference was observed.
Change in blood pressure | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in systolic and diastolic blood pressure was observed.
Change in glycated hemoglobin | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in glycated hemoglobin was observed.
Change in glucose level | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in glucose level was observed.
Change in LDL-cholesterol | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in LDL-cholesterol level was observed.
Change in aspartate transaminase (AST) level | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in aspartate transaminase (AST) level was observed.
Change in antioxidant potential of serum | 12 weeks
  After 8 weeks of using chokeberry juice-100 mL daily and another 4 weeks of using chokeberry juice - 100 mL daily and chokeberry fiber - 10 g daily, a change in antioxidant potential of serum was observed.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata E. Zujko, Dr., Principal Investigator — Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Undecided